CLINICAL TRIAL: NCT01749982
Title: A Pilot Study of Choline and Betaine Supplementation in Arsenic-exposed Individuals in Bangladesh
Brief Title: A Preliminary Study of Choline and Betaine Supplementation Among Adults Exposed to Arsenic in Bangladesh
Acronym: CABS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Megan Hall, Assistant Professor of Epidemiology, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: AAAJ1959
Record Dates: First submitted 2012-12-12; First posted 2012-12-17 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Arsenic Metabolites Measured in Urine
Keywords: arsenic; Bangladesh; choline; betaine; methylation
MeSH Terms: interventions — Choline; Betaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo tablets
  Interventions: Other: Placebo
- Choline bitartrate (Experimental): Choline bitartrate 700 mg by mouth daily
  Interventions: Drug: Choline bitartrate
- Betaine (Experimental): Betaine 1000 mg by mouth daily
  Interventions: Drug: Betaine
- Choline bitartrate + Betaine (Experimental): Choline bitartrate 700 mg + Betaine 1000 mg daily
  Interventions: Drug: Choline bitartrate + Betaine

INTERVENTIONS:
Other: Placebo
  Arms: Placebo
Drug: Choline bitartrate
  Arms: Choline bitartrate
Drug: Betaine
  Arms: Betaine
Drug: Choline bitartrate + Betaine
  Arms: Choline bitartrate + Betaine

SUMMARY:
Roughly 140 million people worldwide are chronically exposed to As-contaminated drinking water at concentrations exceeding the World Health Organization (WHO) standard of 10 µg/L. Arsenic is a class I carcinogen known to cause several types of cancer and ischemic heart disease. Metabolism of inorganic As (InAs), which facilitates urinary As excretion, relies on one-carbon metabolism and involves two methylation steps; both utilize S-adenosylmethionine (SAM) as the methyl donor. SAM biosynthesis relies on B vitamins including folate and B12 for the recruitment and transfer of methyl groups, but other nutrients, including choline and betaine, also contribute to the methyl pool. Our recent findings from a cross-sectional study of Bangladeshi adults exposed to a wide range of As concentrations in drinking water show that plasma choline and betaine concentrations are positively associated with As methylation. These findings suggest that choline and/or betaine may play an important role in As methylation and elimination and that simple interventions may have therapeutic potential for the many populations at risk for As-induced health effects.

The investigators aim to recruit and follow 60 participants for this pilot study which will allow us to 1) assess the acceptance of choline and betaine supplements, 2) monitor participants for any potential side effects, 3) identify any difficulties that might be encountered in daily follow-up, and 4) generate preliminary data regarding the effects of choline and/or betaine supplementation on arsenic methylation.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65
* Absence of all exclusion criteria

Exclusion Criteria:

* women who are currently pregnant at the time of recruitment and/or plan to become pregnant within 2 months
* individuals taking nutritional supplements at the time of recruitment
* individuals who have taken nutritional supplements within the last 3 months
* participants enrolled in any other clinical trial
* women who are currently breastfeeding
* individuals known to have coronary heart disease, cerebrovascular disease, hypertension, renal disease, chronic obstructive pulmonary disease, asthma, cancer, or liver disease
* participants with protein or glucose in their urine sample (dipstick test)
* individuals whose drinking water history is complete for < 3 months

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan N Hall, ScD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Arsenic Research Project, Dhaka, Bangladesh

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo tablets
  Placebo
- Choline Bitartrate: Choline bitartrate 700 mg by mouth daily
  Choline bitartrate
- Betaine: Betaine 1000 mg by mouth daily
  Betaine
- Choline Bitartrate + Betaine: Choline bitartrate 700 mg + Betaine 1000 mg daily
  Choline bitartrate + Betaine
Period: Overall Study
Arm/Group | Placebo | Choline Bitartrate | Betaine | Choline Bitartrate + Betaine
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 12
Not Completed | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Choline Bitartrate | Betaine | Choline Bitartrate + Betaine | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Customized [Median (Full Range); unit: years] | 30.0 [21.0 to 42.0] | 34.0 [25.0 to 43.0] | 29.0 [25.0 to 45.0] | 32.0 [20.0 to 48.0] | 31.0 [21 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 7 | 30
  Male | 7 | 7 | 8 | 8 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 15 | 15 | 15 | 15 | 60
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 15 | 15 | 15 | 15 | 60
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Bangladesh | 15 | 15 | 15 | 15 | 60

OUTCOME MEASURES:

1. Primary Outcome: Change in Urinary % Monomethyl Arsenic
Time Frame: From baseline to 8 weeks after the start of the intervention (week 8 - baseline)
Measure: Median (Full Range); unit: percentage of total urinary arsenic
Arm/Group | Placebo | Choline Bitartrate | Betaine | Choline Bitartrate + Betaine
Number analyzed (Participants) | 15 | 15 | 15 | 12
percentage of total urinary arsenic | 2.4 [-8.4 to 7.8] | 0.24 [-4.3 to 9.4] | -0.06 [-11.6 to 5.4] | -3.2 [-8.9 to 1.2]

2. Primary Outcome: Change in Urinary % Inorganic Arsenic
Time Frame: From baseline to 8 weeks after the start of the intervention (week 8 - baseline)
Measure: Median (Full Range); unit: percentage of total urinary arsenic
Arm/Group | Placebo | Choline Bitartrate | Betaine | Choline Bitartrate + Betaine
Number analyzed (Participants) | 15 | 15 | 15 | 12
percentage of total urinary arsenic | 3.0 [-13.2 to 10.3] | -0.87 [-21.7 to 20.8] | -1.25 [-8.2 to 8.2] | -1.7 [-12.7 to 26.7]

3. Primary Outcome: Change in Urinary % Dimethyl Arsenic
Time Frame: From baseline to 8 weeks after the start of the intervention (week 8 - baseline)
Measure: Median (Full Range); unit: percentage of total urinary arsenic
Arm/Group | Placebo | Choline Bitartrate | Betaine | Choline Bitartrate + Betaine
Number analyzed (Participants) | 15 | 15 | 15 | 12
percentage of total urinary arsenic | -5.8 [-11.5 to 21.6] | 0.65 [-16.4 to 15.3] | -0.87 [-13.4 to 13.9] | 5.45 [-20.8 to 18.5]

ADVERSE EVENTS:
Arm/Group | Placebo | Choline Bitartrate | Betaine | Choline Bitartrate + Betaine
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 5/15 | 5/15 | 2/15 | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Choline Bitartrate (N=15) | Betaine (N=15) | Choline Bitartrate + Betaine (N=15)
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 0 | 2
Fever (General disorders) | 3 | 2 | 2 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
This is a pilot study that is not powered to detect statistically significant effects. The results given here are descriptive.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No